CLINICAL TRIAL: NCT06562842
Title: The Effects of Regular Exercise on Gut Microbiota Composition in Individuals with Type 2 Diabetes
Brief Title: Exercise, Gut Microbiota and Type 2 Diabetes
Acronym: Ex-GM-T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Ex-GM-T2D study
Record Dates: First submitted 2024-08-10; First posted 2024-08-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- NGT - Exercise (Experimental): Regular exercise for 12 weeks and detraining for 4 weeks
  Interventions: Other: Regular exercise
- NGT - Control comparator (Active Comparator): Sedentary behavior for 16 weeks
  Interventions: Other: Control comparator
- Pre-D - Exercise (Experimental): Regular exercise for 12 weeks and detraining for 4 weeks
  Interventions: Other: Regular exercise
- Pre-D - Control comparator (Active Comparator): Sedentary behavior for 16 weeks
  Interventions: Other: Control comparator
- T2D - Exercise (Experimental): Regular exercise for 12 weeks and detraining for 4 weeks
  Interventions: Other: Regular exercise
- T2D - Control comparator (Active Comparator): Sedentary behavior for 16 weeks
  Interventions: Other: Control comparator

INTERVENTIONS:
Other: Regular exercise — Participants will perform regular exercise training for 12 weeks, followed by 4 weeks of detraining.
  Arms: NGT - Exercise; Pre-D - Exercise; T2D - Exercise
Other: Control comparator — Participants will remain sedentary throughout the 16-weeks intervention period.
  Arms: NGT - Control comparator; Pre-D - Control comparator; T2D - Control comparator

SUMMARY:
This randomized, parallel, controlled study, will investigate the effect of regular exercise on GM composition, inflammatory status, and insulin sensitivity, in the progression from normal glucose tolerance (NGT), to prediabetes (pre-D), to type 2 diabetes (T2D). Following baseline assessment of glucose tolerance, the participants will be randomly assigned to either a 12-week, thrice-weekly exercise training program followed by 4 weeks of detraining, or will remain sedentary for the 16-week intervention. Thus, the six study groups will be: 1) NGT group (NGT), NGT individuals - no exercise, 2) NGT exercise group (NGT+Ex), NGT individuals that will participate in training and detraining, 3) pre-D group (pre-D), pre-D individuals - no exercise, 4) pre-D exercise group (Pre-D+Ex), pre-D individuals that will participate in training and detraining, 5) T2D group (T2D), T2D individuals - no exercise, and 6) T2D exercise group (T2D+Ex), T2D individuals that will participate in training and detraining. Assessment of physiological measures, anthropometric characteristics, body composition, glucose tolerance, insulin sensitivity, complete blood count, lipidemic profile, GM composition, inflammatory status, oxidative stress, and muscle performance, will be conducted before and following 12 weeks of the exercise training intervention and following 4 weeks of detraining for all participants.

DETAILED DESCRIPTION:
Type 2 diabetes is a global metabolic epidemic and a major global health threat. In 2021, 537 million adults aged 20-79 years worldwide had diabetes. T2D, is related with life threatening microvascular and macrovascular health complications that contribute tremendously to the burden of mortality and disability worldwide. T2D is defined by fasting hyperglycemia which is largely secondary to inadequate action of insulin. T2D is usually preceded by a state of intermediate hyperglycemia or Pre-D, which is characterized by impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both, and greatly increases the risk for T2D. In T2D, although insulin levels are normal or high, tissues such as liver, skeletal muscle, and adipose tissue become resistant to insulin resulting in high levels of blood glucose. T2D is associated with a systemic inflammatory response which seems to be an independent risk factor for the development of T2D. Additionally, individuals with T2D tend to have a more oxidative internal environment than healthy subjects. Hyperglycemia-induced oxidative stress has been found to affect the insulin signaling cascade and decrease GLUT4 gene transcription and also alter mitochondrial activity. T2D pathophysiology has also been associated with GM composition. Dysbiosis of GM is suggested to have a central role in the pathogenesis of insulin resistance and T2D through several mechanisms.

The important role of regular exercise for the prevention and treatment of T2D has been established. Most benefits of exercise on T2D management and prevention are realized through the adaptations to skeletal muscle which in turn induce acute and chronic improvements in insulin action. Exercise also exerts anti-inflammatory effects. Emerged evidence suggests that exercise may also favorably affect T2D by improving GM composition. The most promising effect of regular exercise is the alteration of GM towards a healthier microbial composition by producing a more diverse GM, decreasing pathogenic bacterial communities and increasing SCFAs-producing bacteria. However, the impact of exercise on the GM structure and function of T2D individuals is poorly understood, as only a limited number of studies exist in this area, so far.

According to a preliminary power analysis (a probability error of 0.05 and a statistical power of 80%), a sample size of 8-10 participants/group was considered appropriate to detect statistically meaningful changes between trials. Thus, ≥60 middle-aged individuals will be assessed for eligibility to participate in the study. The study will be conducted in a parallel, randomized, controlled design. The participants, will be primarily informed of the study procedures, as well as the benefits and possible risks, and they will also sign an informed consent form for participation in the study. All eligible individuals will provide blood samples for the determination of fasting blood glucose, glycosylated hemoglobin (HbA1c), and fasting plasma insulin, and will take an oral glucose tolerance test (OGTT) to determine their glycemic profile, according to which, they will be characterized as normal glucose tolerance (NGT) individuals, or pre-diabetes (pre-D) individuals, or type 2 diabetes (T2D) individuals. Physical activity levels will also be assessed through the International Physical Activity Questionnaire (IPAQ). Afterwards, the participants of each glucose tolerance stage will be randomly assigned to either the 12 weeks of regular combined aerobic and resistance exercise according to the guidelines for pre-D and T2D individuals, or remain sedentary for 12 weeks. Thus, six intervention groups will be as follows: i) NGT group (NGTG), NGT individuals - no exercise, ii) NGT exercise group (NGTG+Ex), NGT individuals that will participate in training and detraining, iii) pre-D group (pre-DG), pre-D individuals - no exercise, iv) pre-D exercise group (Pre-DG+Ex), pre-D individuals that will participate in training and detraining, v) T2D group (T2DG), T2D individuals - no exercise, and vi) T2D exercise group (T2DG+Ex), T2D individuals that will participate in training and detraining. Randomization of the conditions will be done by a software generating random integers available on the internet (Random.org).

Baseline measurements will take place at the Laboratory of Biochemistry, Physiology and Nutrition of Exercise (SmArT Lab), Department of Physical Education and Sports, University of Thessaly: physiological measures (resting heart rate, resting systolic and diastolic blood pressure, resting metabolic rate), anthropometric characteristics (body height, body mass, body mass index), body composition (amount of body fat, lean body mass, fat mass, bone density), muscle performance [aerobic capacity (VO2max), isokinetic strength of the lower extremities (isometric, concentric and eccentric torque of the knee extensors and knee flexors), handgrip strength, muscle power (countermovement jump)]. Additionally, the participants will provide feces for the determination of GM composition and GM metabolites [short chain fatty acids (SCFAs)], as well as blood samples for the determination of complete blood count (CBC), systemic inflammation [tumor necrosis factor alpha (TNF-α), interleukin 6 (IL-6), C-reactive protein (CRP), zonulin, lipopolysaccharides-binding protein (LBP)], blood redox status [total antioxidant capacity (TAC), catalase (CAT), protein carbonyls (PC), reduced glutathione (GSH), oxidized glutathione (GSSG), GSH/GSSG ratio, malondialdehyde (MDA), uric acid, bilirubin], and lipid profile [total cholesterol (CHO-T), low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides (TG)]. In addition, the participants will record their diet via a 7-days recall before their participation in the first experimental condition, and dietary data will be analyzed. All of the above measurements will be repeated following the 12-weeks of exercise intervention, as well as following the 4-weeks of detraining period. The participants that will be allocated into the regular exercise, except for VO2max, they will further undergo estimation of maximal strength of the main muscle groups for the determination of intensity of each participant's exercise program; aerobic capacity and muscle strength determination will also be repeated after four weeks of the regular exercise for the necessary intensity adjustments of the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years old
* Sedentary lifestyle or insufficient daily physical activity according to guidelines for T2D
* Abstinence of anti-inflammatory drugs and/or antibiotics and/or dietary supplements that could affect GM composition before the study (>3 months)
* No other chronic diseases and/or musculoskeletal injuries (>6 months)

Exclusion Criteria:

* Age <45 years or >65 years
* Physically active individuals
* Consumption of anti-inflammatory drugs and/or antibiotics and/or dietary supplements that could affect GM composition before the study (<3 months)
* Other chronic diseases ot recent history of musculoskeletal injury (<6 months)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Gut microbiota composition will be assessed in feces via Next generation sequencing
Changes in butyrate | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Butyrate will be assessed in feces via HPLC/MS
Changes in propionate | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Propionate will be assessed in feces via HPLC/MS
Changes in acetate | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Acetate will be assessed in feces via HPLC/MS
Changes in White blood cells (WBC) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  WBC will be assessed in whole blood via hematological analyzer
Changes in Lymphocytes (LYM) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  LYM will be assessed in whole blood via hematological analyzer
Changes in Monocytes (MON) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MON will be assessed in whole blood via hematological analyzer
Changes in Granulocytes (GRA) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  GRA will be assessed in whole blood via hematological analyzer
Changes in percent Lymphocytes (LYM%) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  LYM% will be assessed in whole blood via hematological analyzer
Changes in percent Monocytes (MON%) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MON% will be assessed in whole blood via hematological analyzer
Changes in percent Granulocytes (GRA%) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  GRA% will be assessed in whole blood via hematological analyzer
Changes in Red blood cells (RBC) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  RBC will be assessed in whole blood via hematological analyzer
Changes in Hemoglobin (HGB) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  HGB will be assessed in whole blood via hematological analyzer
Changes in Hematocrit (HCT) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  HCT will be assessed in whole blood via hematological analyzer
Changes in Mean corpuscular volume (MCV) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MCV will be assessed in whole blood via hematological analyzer
Changes in Mean corpuscular hemoglobin (MCH) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MCH will be assessed in whole blood via hematological analyzer
Changes in Mean corpuscular hemoglobin concentration (MCHC) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MCHC will be assessed in whole blood via hematological analyzer
Changes in Red cell distribution width (RDW) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  RDW will be assessed in whole blood via hematological analyzer
Changes in Platelets (PLT) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  PLT will be assessed in whole blood via hematological analyzer
Changes in Mean platelets volume (MPV) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MPV will be assessed in whole blood via hematological analyzer
Changes in Plateletcrit (PCT) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  PCT will be assessed in whole blood via hematological analyzer
Changes in Plateletcrit distribution width (PDW) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  PDW will be assessed in whole blood via hematological analyzer
Changes in TNF-α concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  TNF-α concentration will be assessed in serum via ELISA
Changes in IL-6 concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  IL-6 concentration will be assessed in serum via ELISA
Changes in high-sensitivity C-reactive protein concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  C-reactive protein concentration will be assessed in serum via ELISA
Changes in lipopolysacharides-binding protein (LBP) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  LBP concentration will be assessed in serum via ELISA
Changes in zonulin concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Zonulin concentration will be assessed in serum and in feces via ELISA
Changes in protein carbonyls (PC) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  PC concentration will be assessed in plasma via a spectrophotometer
Changes in malondialdehyde (MDA) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  MDA concentration will be assessed in plasma via HPLC
Changes in reduced glutathione (GSH) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  GSH concentration will be assessed in red blood cells lycate via a spectrophotometer
Changes in oxidized glutathione (GSSG) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  GSSG concentration will be assessed in red blood cells lycate via a spectrophotometer
Changes in GSH/GSSG ratio | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  GSH/GSSG ratio will be calculated by dividing GSH concentration with GSSG concentration
Changes in catalase concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Catalase concentration will be assessed in red blood cells lycate via a spectrophotometer
Changes in total antioxidant capacity (TAC) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  TAC will be assessed in red blood cells lycate via a spectrophotometer
Changes in uric acid concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Uric acid concentration will be assessed in serum via a biochemical analyzer
Changes in bilirubin concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Bilirubin concentration will be assessed in serum via a biochemical analyzer
Changes in glycosylated hemoblobin (HbA1c) concentration | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  HbA1c concentration will be assessed in whole blood via a HbA1c analyzer
Changes in fasting plasma glucose | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Fasting plasma glucose will be assessed in plasma via a biochemical analyzer
Changes in fasting plasma insulin | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Fasting plasma insulin will be assessed in plasma via a biochemical analyzer
Changes in insulin resistance | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Insulin resistance will be calulated via the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) index
Changes in insulin resistance - Oral glucose tolerance test (OGTT) | Pre, 30 minutes post-, 60 minutes post-, 90 minutes post-,120 minutes post-glucose consumption
  OGTT will be assessed via the estimation of 2-h plasma glucose following oral glucose consumption
Changes in total cholesterol (CHOL-T) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  CHOL-T will be assessed via a biochemical analyzer
Changes in low-density lipoprotein cholesterol (LDL-C) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  LDL-C will be assessed via a biochemical analyzer
Changes in high-density lipoprotein cholesterol (HDL-C) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  HDL-C will be assessed via a biochemical analyzer
Changes in triglycerides (TG) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  TG will be assessed via a biochemical analyzer
Changes in countermovement jump height (CMJ) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  CMJ height will be measured via an optical system
Changes in isokinetic strength of knee extensors and knee flexors | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Isometric, concentric and eccentric peak torque of the knee extensors and knee flexors of both limbs will be assessed via an isokinetic dynamometer
Changes in handgrip strength | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Handgrip strength will be assessed via a handgrip dynamometer
Changes in resting heart rate (HR) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Resting HR will be assessed via a HR monitor
Changes in resting systolic (SBP) and diastolic blood pressure (DBP) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Resting SBP and DBP will be assessed via a manual sphygmomanometer
Changes in resting metabolic rate (RMR) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  RMR will be assessed via indirect calorimetry
Changes in body mass (BM) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  BM will be assessed via a stadiometer-Beam balance
Changes in body height | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Body height will be assessed via a stadiometer-Beam balance
Changes in body mass index (BMI) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  BMI will be calculated by dividing body mass by the square of body height
Changes in maximal oxygen uptake (VO2max) | Baseline (pre), 12 weeks post-training, 16 weeks (post-detraining)
  Changes in maximal oxygen uptake (VO2peak) will be assesed via a submaximal test on a treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K. Deli, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, Uninersity of Thessaly, Trikala, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Gurung M, Li Z, You H, Rodrigues R, Jump DB, Morgun A, Shulzhenko N. Role of gut microbiota in type 2 diabetes pathophysiology. EBioMedicine. 2020 Jan;51:102590. doi: 10.1016/j.ebiom.2019.11.051. Epub 2020 Jan 3. PMID 31901868
- [Background] Pasini E, Corsetti G, Assanelli D, Testa C, Romano C, Dioguardi FS, Aquilani R. Effects of chronic exercise on gut microbiota and intestinal barrier in human with type 2 diabetes. Minerva Med. 2019 Feb;110(1):3-11. doi: 10.23736/S0026-4806.18.05589-1. PMID 30667205
- [Background] Torquati L, Gajanand T, Cox ER, Willis CRG, Zaugg J, Keating SE, Coombes JS. Effects of exercise intensity on gut microbiome composition and function in people with type 2 diabetes. Eur J Sport Sci. 2023 Apr;23(4):530-541. doi: 10.1080/17461391.2022.2035436. Epub 2022 Mar 23. PMID 35107058